CLINICAL TRIAL: NCT05482074
Title: Pilot Trial of Olaparib in Patients With Unresectable or Metastatic Melanoma With Mutations in BRCA1/2 Genes
Brief Title: Olaparib in Unresectable/Metastatic Melanoma With BRCA1/2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left the institute
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-294
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Recurrent Metastatic Melanoma; Cutaneous Melanoma; Mucosal Melanoma; Uveal Melanoma
Keywords: Recurrent metastatic melanoma; Cutaneous Melanoma; Mucosal Melanoma; Uveal Melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OLAPARIB (Experimental): The research study procedures include screening for eligibility, study treatment including evaluations, surveys, optional biopsies, and follow up visits
  Olaparib- Each study treatment cycle lasts 28 days . This will continue for as long as the study treatment is providing clinical benefit
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Oral, twice a day, dosage per protocol, per 28 day cycle
  Other Names: LYNPARZA

SUMMARY:
The purpose of this study is to evaluate how effective Olaparib is when given as a treatment for primary or recurrent, unresectable or metastatic melanoma. This research study involves targeted therapy.

-The name of the study drug involved in this study is: Olaparib (also known as Lynparza)

DETAILED DESCRIPTION:
A phase II, single arm, open label pilot trial in a sample size of 15 primary or recurrent, unresectable or metastatic melanoma patients that have progressed on prior checkpoint inhibitor therapy with germline or somatic mutations in BRCA1/2.

The research study procedures include screening for eligibility, study treatment including evaluations, surveys, optional biopsies, and follow up visits. This research study involves targeted therapy.

* The name of the study drug involved in this study is:
* Olaparib (also known as Lynparza)

It is expected that about 15 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

This research study is a Pilot Study, which is the first time investigators are examining this drug for treatment of melanoma.

The U.S. Food and Drug Administration (FDA) has not approved Olaparib for this specific disease, but it has been approved for other uses.

AstraZeneca, a pharmaceutical company, is supporting this research study by providing funding for the research study and the study drug, Olaparib.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed diagnosis of primary or recurrent metastatic melanoma including cutaneous, mucosal, or uveal melanoma.
* Participants must have a germline or somatic DNA damage repair mutation or deletion in BRCA1 or BRCA2. The result may have been obtained from one of the following test providers: OncoPanel, SNaPshot Panel, Myriad Genetics, Invitae, Ambry, Quest, Colour Genomics, IMPACT, Foundation Medicine (tissue or ctDNA based), Guardant, or another CLIA approved tissue and/or serum based next generation sequencing-based assay. (Variants of uncertain significance are excluded.)
* Participants must have measurable disease as defined by RECIST 1.1 criteria

  * At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) (or Clinical examination) and which is suitable for accurate repeated measurements.
  * Subjects must have received prior checkpoint inhibitor therapy (defined as anti-CTLA4 or anti-PD-1 or combination anti-CTLA4/anti-PD-1), either for metastatic or unresectable disease or progressed on adjuvant therapy.
  * Age ≥18 years. Because no dosing or adverse event data are currently available on the use of olaparib in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Patients must have a life expectancy ≥ 16 weeks.
* ECOG performance status ≤1(Karnofsky ≥60%, see Appendix A).
* Participants must have adequate organ and marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
  * Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test: Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)a / serum creatinine (mg/dL) x 72 (where F=0.85 for females and F=1 for males).
* Participants must have the ability to swallow pills.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The effects of olaparib on the developing human fetus are unknown. For this reason and because similar agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.
* Postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
  * radiation-induced oophorectomy with last menses >1 year ago
  * chemotherapy-induced menopause with >1 year interval since last menses
  * surgical sterilization (bilateral oophorectomy or hysterectomy)
* Measurable disease as defined by RECIST 1.1 criteria

  -- At least one lesion, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) (or Clinical examination) and which is suitable for accurate repeated measurements.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy (except for palliative reasons) for melanoma within 3 weeks prior to entering the study.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities CTCAE > Grade 2) with the exception of alopecia.
* Participants who are receiving any other investigational agents.
* Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma. Patients with a history of localized triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
* Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Any previous treatment with a PARP inhibitor, including olaparib.
* Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because olaparib is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib breastfeeding should be discontinued if the mother is treated with olaparib.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Known HIV or AIDS-related illness.
* Patients with known active hepatitis (i.e. Hepatitis B or C).

  * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-04 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 12 weeks
  Best overall response (CR+PR) assessed by RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival | from first dose of treatment until disease progression or death up to 2 years
  assessed by RECIST v1.1
Number of participants with treatment-related adverse events | from first dose of treatment up to 2 years
  NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0,
Disease Control Rate | start of treatment until disease progression up to 2 years
  (Complete Response+ Partial Response + Stable Disease) by RECIST v1.1
Overall Survival | defined as the time from start of treatment to the date of death due to any cause up to 5 Years
  Time from start of treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Sussman, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu